CLINICAL TRIAL: NCT05721703
Title: Observe the Multi-indices of Long-term Peritoneal Dialysis Patients to Explore the Evolution of Peritoneal Ultrafiltration Failure
Brief Title: An Observational Study of Long-term Peritoneal Dialysis Patients Who Eventually Develop Ultrafiltration Failure (LUFF)
Acronym: LUFF
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jianhui Zhou, Director, Blood purification Branch, Division of Nephrology, Principal Investigator, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: S2021-263-01
Record Dates: First submitted 2022-10-04; First posted 2023-02-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Ultrafiltration Failure
Keywords: peritoneal dialysis; Ultrafiltration Failure; long-term

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood, dialysate, etc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
At present, there are few researches on peritoneal dialysis, especially on ultrafiltration failure of peritoneal dialysis. To explore the regularity and mechanism of peritoneal ultrafiltration failure,investigators followed up the comprehensive data of participants from the insertion to the removal of the peritoneal dialysis catheter, and collected the peritoneal tissue for morphological and single-cell analysis when the participants inserting or removing their catheters. If the catheter is still in use when this study stop collecting data, the peritoneal dialysis effluent will substitute for peritoneal tissue to the morphological and single-cell analysis. Clinical data and single-cell sequence data were processed using statistical analyses to identify factors affecting ultrafiltration failure.

DETAILED DESCRIPTION:
Background: Chronic kidney disease (CKD) is one of the most common non-communicable diseases. The Global Burden of Disease (GBD), which examined multiple diseases in 188 countries from 1990 to 2013, found that the number of CKD patients increased from 318,665,000 to 47,1916,000, representing a 48% increase in prevalence (2.1% annually). Peritoneal dialysis is an important renal replacement therapy for participants with end-stage renal disease. The removal of water mainly depends on the high osmotic pressure of dialysate which is called ultrafiltration, and the loss of ultrafiltration function of peritoneum is called ultrafiltration failure. Data from the National Blood Purification Case Information System (CNRDS) show that the rate of conversion from ultrafiltration failure to hemodialysis is 5%-10%, and cardiovascular complications caused by fluid overload, such as malignant hypertension and heart failure, are the common causes of death. At the end of 2021, dialysis data in mainland China showed that there were nearly 880,000 patients undergoing dialysis treatment, of which 14% chose peritoneal dialysis, the average dialysis age of peritoneal dialysis patients was 50.3 months, the proportion of patients who had been on dialysis for more than 5 years was 33.9%, and the proportion of patients who had been on dialysis for more than 10 years was 7.5%. It can be seen that long-term peritoneal dialysis still has a high shedding rate, and ultrafiltration failure is the key problem of long-term peritoneal dialysis.

Methods: Investigators gathered participants from Department of Nephrology, PLA General Hospital, from May 2021 to May 2029. Inclusion Criteria: 1.Clinically diagnosed as chronic renal insufficiency (CKD 5); 2.Incident PD patients who were newly inserted PD catheter during the observation period of this study; 3.Prevalent PD patients who inserted PD cather before initiation of this study, should be admitted as pre-UFF, has taken long-term PD(>5 years) before removing cather during the observation period of this study; 4.Written informed consent signed by the patient or the authorized client has been obtained. Exclusion Criteria: 1.Acute renal failure; 2.Pregnant or lactating women; 3.Active infection duration; 4.One of infectious serum markers of HIV, syphilis, hepatitis B and hepatitis C is positive; 5.Any other conditions that the investigator considers impossible to join this trial. The observed indices were: (1)Demographic characteristics; (2)Peritoneal equilibration test (PET D/P), adequacy assessment(Ccr, Kt/V), evaluation of ultrafiltration (urine volume, intake,etc.); (3)Peritoneal dialysate routine examination, peritoneal dialysate inflammation examination and other markers and exosome examination; (4)Classification and counting of exfoliated cells from peritoneal dialysis effluent, and dialysate exfoliated cells primary culture for further cell biology analysis; (5)Peritoneal histopathology and immunohistochemical analysis and proteomics and single cell transcriptome analysis; (6)Clinical examinations: Routine blood test, Uroscopy, Blood biochemistry test, Coagulation function test, Immunoassay, Bone metabolism test, Thyroid function test, Evaluation of Ascites, etc. For an incident PD patient,after admission，the peritoneal catheter was inserted, and the data of the initial peritoneal equilibration test and clinical examinations were collected, and the peritoneal membrane was sampled for single-cell analysis. After that, the patient was followed up, and the data of the subsequent peritoneal equilibration test and clinical examinations were collected until the end point(technique failure) or the study end(8 years). The investigators collected the peritoneal tissue for single-cell sequencing when participants remove the catheters(for the technique failure patients). If the catheter is still in use when this study stop collecting data(8 years), the peritoneal dialysis effluent will substitute for peritoneal tissue to the morphological and single-cell analysis. For a prevalent patient who admitted as pre-UFF, investigators collected the final peritoneal equilibration test and clinical examination data then sample the peritoneal tissue for single-cell sequencing when removing the cather. SPSS and R were used for statistical analysis. Continuous variables were expressed as mean ± standard deviation, and discontinuous variables were expressed as percentage. The independent t-test or chi-square test was used for comparison between the two data. P<0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed as chronic renal insufficiency (CKD 5)
2. Patients who met the first dialysis guidelines for peritoneal dialysis without catheter, or patients with peritoneal dialysis regularly, or ultrafiltration failure was diagnosed and patients on peritoneal dialysis were to be existed.
3. Written informed consent signed by the patient or the authorized client has been obtained.

Exclusion Criteria:

1. Acute renal failure.
2. Pregnant or lactating women.
3. Active infection duration.
4. One of infectious serum markers of HIV, syphilis, hepatitis B and hepatitis C is positive.
5. Any other conditions that the investigator considers impossible to join this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were diagnosed CKD5 age 18 to 70 need or keep peritoneal dialysis to treat or someone was ultrafiltration failure without AKI, pregnant or lactating women, active infection, infectious diseases and be asked to sign an "informed consent form".
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical survival rate | 8 year
  Technical survival of peritoneal dialysis

SECONDARY OUTCOMES:
D/P | 1,2,3,4,5,6,7,8 year
  Ratio of substance content in peritoneal dialysate to that in blood.
OCG | 1,2,3,4,5,6,7,8 year
  Glucose transport rates measured by a double mini peritoneal equilibration test.
Ccr | 1,2,3,4,5,6,7,8 year
  Creatinine clearance rate. Ccr=urinary creatinine concentration * urine volume per minute/blood creatinine concentration.
Kt/V | 1,2,3,4,5,6,7,8 year
  Ratio of urea clearance to volume during unit dialysis time.
Cell counting | 1,2,3,4,5,6,7,8 year
  Count the number of cells.
Electrolyte | 1,2,3,4,5,6,7,8 year
  Content of ions.
Blood biochemical index | 1,2,3,4,5,6,7,8 year
  Venous blood was obtained for biochemical examination.
Urine protein | 1,2,3,4,5,6,7,8 year
  Urine test for protein content.
Histopathology | 1,2,3,4,5,6,7,8 year
  With the consent of the patients, peritoneal tissue was taken to observe histological changes.
Single-cell transcriptome sequencing | 1,2,3,4,5,6,7,8 year
  With the consent of the patients, tissues were taken for analysis. Isolate cells in the tissues and measure gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: CHEN Xiangmei, yes, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China